CLINICAL TRIAL: NCT04006158
Title: A Controlled Study to Investigate the Effect of a Multi-wave Light Emitting Diode (LED) Bed on Blood Pressure and Endothelial Function
Brief Title: A Controlled Study to Investigate the Effect of Multi-wave Light Emitting Diode (LED) Bed on Blood Pressure and Endothelial Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LED Intellectual Properties, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Light bed hypertension
Record Dates: First submitted 2019-06-29; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- LightStim LED Bed (Experimental): Full body LED bed device.
  Interventions: Device: LED bed

INTERVENTIONS:
Device: LED bed — Low risk FDA cleared full body LED bed

SUMMARY:
The objective of this multi-center study is to investigate the effect of a multi-wave LED light bed on blood pressure and endothelial function in pre-hypertensive and mildly hypertensive adults.

DETAILED DESCRIPTION:
Subjects will be instructed to lay in the bed for 20 minutes on their stomach followed by 20 minutes on their back for a total of 40 minutes three times per week for 8 weeks. Subjects will be instructed to begin light treatment on Day 1 after baseline measurements have been collected. Subjects will be required to visit a Wellness Center of Dr. Bryan or Hypertension Institute in Nashville, informed of the study and if agreed will sign the consent form. After consent, subjects will be required to spend about 30 minutes to get baseline measurements. Subjects will then be required to lie in bed for 40 minutes each day three days per week for 8 weeks. Blood pressure and endothelial function tests will be recorded at baseline and after each light treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of 18-75 years of age
* If female, subject is not of child bearing potential
* Subjects with seated resting systolic blood pressures between 130-160 mmHg and diastolic between 85-100 mmHg (inclusive) at screening visit
* Subjects with mild to moderate endothelial dysfunction
* Agreement to maintain current level of physical activity and diet throughout the study
* Agrees to comply with study procedures including abstain from coffee at least 14 hours before blood pressure measurement and abstain from physical exercise at least 4 hours before blood pressure measurement
* Has given voluntary, written, and informed consent to participate in the study

Exclusion Criteria:

* Females who are pregnant, breastfeeding, or planning to become pregnant during the course of the study
* Seated office systolic blood pressure outside of the target range (systolic blood pressure <130 mmHg or >160 mmHg) or diastolic blood pressure <85 or >100 mmHg at screening
* The use of natural health products for the treatment of hypertension within 2 weeks of screening
* Significant cardiac history defined as a history of myocardial infarction (MI); coronary angioplasty or bypass graft(s); Valvular disease or repair; unstable angina pectoris; transient ischemic attack (TIA); cerebrovascular accidents (CVA); congestive heart failure; or coronary artery disease (CAD)
* Type I diabetes
* Unstable medical conditions that in the opinion of the Principle Investigator preclude the subject from participating in the study
* Alcohol or drug abuse within the last 6 months
* Participation in a clinical research trial within 30 days prior to randomization
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-29 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Hypertension | 8 weeks
  The primary efficacy outcome to be analyzed is the between-group changes from baseline (Day 0) to end of study (Day 60) in daytime mean systolic and diastolic BP and endothelial function, measured using a triplicate readings using AHA guidelines and MaxPulse, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Nitric Oxide Innovations, Rockdale, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided